CLINICAL TRIAL: NCT06663709
Title: Effect of Balance, Resistance, Aerobic, Cognitive Exercises(BRACE)on Balance, Cognition and Mobility Among Stroke Patients
Brief Title: Effect of BRACE on Balance, Cognition and Mobility Among Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Sadia Bashir
Record Dates: First submitted 2024-10-28; First posted 2024-10-29 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Stroke Patients
Keywords: BRACE Protocol; Task Oriented Protocol; Stroke Population; Balance Impairments
MeSH Terms: interventions — Braces

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Balance Resistance Aerobic Cognitive Exercises (BRACE) (Experimental): BRACE include combination of exercises including, Balance, Resistance, Aerobic, Cognition Exercises.
  Interventions: Other: BRACE
- Task Oriented (Experimental): Task Oriented protocol is combination of warm up, balance,,and cognition exercises.
  Interventions: Other: TASK-oriented

INTERVENTIONS:
Other: BRACE — Study will be conducted after the approval of Ethical review board. The BRACE exercise training would be perform in 3 times a week for 9 weeks, lasting approximately 40-60 minutes each time. Week 0-3 : Balance: Romberg, tandem standing, single leg stance TUG test Resistance: chair rise, Stair climbing Aerobic exercises: 6mint walk, count reverse from 30, push wall and reverse count from 20 Cognitive: count reverse from 50. Week 4-6: Balance: Sit to stand, functional reach, Tug Test, Perturbation, Kick a ball Resistance: stair climbing Aerobic Exercises: Marching in space, Cycling Cognitive: Remember 5 words, spell backward, remember 5 animals Week 7-9: Balance: Combination of all Resistance: Combination of all Aerobic Exercises: Cycling , Marching, 6 min Walk Cognitive: Combination of all
  Arms: Balance Resistance Aerobic Cognitive Exercises (BRACE)
Other: TASK-oriented — Study will be conducted after the approval of Ethical review board. Task oriented training would be perform in 3 times a week for 9 weeks, lasting approximately 40-60 minutes each time. Week 1-3 Warm Up (sit to stand,5 reps)(cycling 3-5 min) , Single leg stand with eye open 15 sec, with eye close 10sec, forward, backward, and side stepping (5 reps) reaching, Transition from sit to stand, Walk then back to sit (3 min),Walk with even steps(3min) Walk with carrying objects. (3min) Week 4-6 Warm up Period, Task oriented training (7 Reps of each task) Week 7-9 Warm up Period, Task oriented training (9Reps of each task)
  Arms: Task Oriented

SUMMARY:
The Objective of the is to determine effect of balance, resistance, aerobic, cognitive exercises (BRACE) protocol on balance, cognition and mobility among stroke patients and to compare the effect of Balance, Resistance, Aerobic, and Cognitive Exercise (BRACE) and task-oriented training on balance cognition and mobility in stroke patients. The study will be randomized control trial including 2 experimental groups with estimated 21 individual in each group.

DETAILED DESCRIPTION:
Stroke is a major and growing global health concern. According to the most current estimates of the Global Burden of Disease (GBD) (2019) stroke burden, stroke continues to be the world's second-leading cause of death and the third-leading cause of death and disability. Stroke is the second most prevalent cause of disability worldwide, and survivors frequently experience impairments to their hands and cognitive functions. Because strokes and sudden cerebrovascular accidents occur so often and have such fatal effects, they remain among the most dangerous global health concerns.

Generally, stroke patients experience diminished motor abilities, as well as impairments to their senses, cognition, and visual perception. In addition, they experience compromised physical function, which makes walking independently challenging because of reduced gait endurance, speed of walking, and balance. Patients with such a decrease in their ability to maintain balance find challenging to walk and perform useful movements, which can cause problems in day-to-day living. Moreover, a stroke patient's ability to walk may be even worse if they fall.

Another major cause of stress for survivors of stroke is the cognitive effect, since they may experience issues with concentration, working memory, and remembering.

Trunk function impairments tend to occur in survivors of strokes. Impaired center of pressure control when sitting, muscular weakness and prolonged trunk muscle activation, severe errors in trunk position awareness, poor trunk performance, and trunk imbalance during walking have all been documented in prior research.

Rehabilitative treatment is a particularly effective therapy in terms of improving recovery from impairment. The objective of rehabilitation is "to achieve and sustain maximum performance in the emotional, mental, and physical domains" .A greater awareness of the neurological underpinnings of therapeutic restoration has occurred with a greater awareness of the former.

Numerous publications that focus on balancing training exercises, strength exercises, and aerobic activities independently have been published in the past several years. BRACE, which stands for Balance, Resistance, Aerobic, and Cognition Exercises, is a new treatment protocol meant to reduce fall risk and improve mobility in older adults. There has not been much work done on the BRACE procedure, therefore we will be focusing on it in this study. Our research compares how Balance Resistance Aerobic Cognitive Exercises (BRACE) affect stroke patients' balance, cognition, and mobility.

ELIGIBILITY:
Inclusion Criteria:

* Hemiplegic stroke patients
* Both genders
* Age:30-65years
* ischemic and hemorrhagic stroke patients
* Sub-acute and chronic patients
* Balance impairment with Berg Balance Scale (BBS) Scores 41-56 score between 18-25 on MoCA (mild cognitive impairment)

Exclusion Criteria:

* Patients who are not willing
* Patients with vision and hearing issue
* A history of serious or unstable cardiac condition
* Orthopedic injuries that could impair locomotion
* History of fall

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2024-10-24 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
Berg And Balance scale | 9 weeks
  changes from the baseline, Berg balance scale (BBS) is used for assessment of balance and fall risk, Higher scores on the BBS indicate greater independence and better ability to balance. In contrast, lower scores indicate a greater fall risk Items DESCRIPTION SCORE (0-4) Sitting to standing, Standing unsupported, Sitting unsupported, Standing to sitting, Transfers , Standing with eyes closed , Standing with feet together, Reaching forward with outstretched arm, Retrieving object from floor, Turning to look behind, Turning 360 degrees, Placing alternate foot on stool, Standing with one foot in front, Standing on one foot, TOTAL __/56
Time Up And Go | 9 weeks
  changes from the baseline, Timed up and go test is used for the assessment of falls risk among the elderly population. The Timed "Up and Go" (TUG) Test measures, in seconds, the time is taken by an individual to stand up from a standard armchair (approximate seat height of 46 cm, arm height 65 cm), walk a distance of 3 meters (approximately 10 feet), turn, walk back to the chair, and sit down. Normal healthy elderly usually complete the task in 10 seconds or less. Very frail or weak elderly with poor mobility may take 2 minutes or more. Clinical guide: <10 seconds = normal <20 seconds = good mobility, can go out alone, mobile without a gait aid <30 seconds = problems, cannot go outside alone, requires a gait aid A score of more than or equal to 14 seconds has been shown to indicate a high risk of falls.
MOCA | 9 weeks
  The Montreal Cognitive Assessment (MOCA) is a cognitive screening instrument developed to detect mild cognitive impairment (MCI). It is a simple 10 min paper and pencil test that assesses multiple cognitive domains including memory, language, executive functions, visuo-patial skills, calculation, abstraction, attention, concentration, and orientation.
  Scores on the MoCA range from zero to 30. A score of 26 and higher is considered normal.
  In the initial study data, normal controls had an average score of 27.4. People with mild cognitive impairment (MCI) scored an average of 22.1. People with Alzheimer's disease had an average score of 16.2.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Azhar, MS-NMPT, Principal Investigator — Riphah International University
Locations (1):
- NIRM, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sherin A, Ul-Haq Z, Fazid S, Shah BH, Khattak MI, Nabi F. Prevalence of stroke in Pakistan: Findings from Khyber Pakhtunkhwa integrated population health survey (KP-IPHS) 2016-17. Pak J Med Sci. 2020 Nov-Dec;36(7):1435-1440. doi: 10.12669/pjms.36.7.2824. PMID 33235553
- [Background] Khallaf ME. Effect of Task-Specific Training on Trunk Control and Balance in Patients with Subacute Stroke. Neurol Res Int. 2020 Nov 17;2020:5090193. doi: 10.1155/2020/5090193. eCollection 2020. PMID 33294224